CLINICAL TRIAL: NCT02463552
Title: Rior Use of Naproxen on Tooth Sensitivity Reduction After In-office Bleaching: Randomized Clinical Trial
Brief Title: Naproxen on Tooth Sensitivity Caused by In-office Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sergipe (Other)
Responsible Party: Principal Investigator, André Luis Faria e Silva, Dr., Universidade Federal de Sergipe
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UFSergipe
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Toothache; Tooth Bleaching
MeSH Terms: conditions — Toothache | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Naproxen
- Naproxen (Experimental)
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — The patient will receive a single-dose of Naproxen (500 mg) one hour before the bleaching procedure.

SUMMARY:
This study aims to evaluate the effects of prior use of non-steroidal anti-inflammatory Naproxen on risk and level of tooth sensitivity caused by in-office bleaching procedures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old patients of both genders presenting good general/oral health;
* All maxillary anterior teeth presenting shade equal or darker than 2M2 at Vita bleachguide guide (Vita-Zahnfabrik, Germany);
* Signed the form accepting to participate of this study.

Exclusion Criteria:

* Presence of caries lesions, restorations and/or endodontic treatment at any maxillary anterior teeth.
* Undergone tooth-whitening procedures;
* Pregnant/lactating;
* Presence of periodontal diseases;
* Presence of severe tooth discoloration by tetracycline stains or fluorosis;
* Any kind of medicine, bruxism habits or any other pathology that can cause sensitivity (such as recession, dentin exposure);
* Continuous use of drugs with anti-inflammatory actions;
* Presence of tooth hypersensitivity at baseline measurement;
* Any known adverse effects caused by Naproxen;
* Non-attendance to any session of evaluation or bleaching.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Risk to Tooth sensitivity - during procedure | During the bleaching procedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Level of tooth sensitivity - during procedure | During the bleaching procedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe.
Risk of tooth sensitivity - after procedure | 24 hours after bleaching prcedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Level of tooth sensitivity - after procedure | 24 hours after bleaching prcedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe.

OTHER OUTCOMES:
Efficacy of bleaching | 7 days after bleaching procedure
  A spectrophotometer will be used to assess the color alteration, while the parameter "L", "a" and "b" will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sergipe, Aracaju, Sergipe, Brazil